CLINICAL TRIAL: NCT05488470
Title: Monitoring QT Intervals Using LINQ/LINQII in Patients Undergoing Antiarrhythmic Drug Loading
Brief Title: QT Changes as Detected From LINQ ECG During Antiarrhythmic Loading (LINQ QT)
Acronym: LINQ QT
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT22018
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-09

CONDITIONS: Atrial Arrhythmia; QT Interval, Variation in; Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: LINQ/LINQ II — Algorithm developed and validated to continuously measure QT intervals for every beat using LINQ/LINQ II ECG. This study is aimed at determining if QT interval changes can be detected during antiarrhythmic drug loading by the designed QT detection algorithm from LINQ/LINQ II ECG.

SUMMARY:
The LINQ QT Study is a prospective, non-randomized, multi-center, observational, post-market clinical study investigating QT interval changes due to antiarrhythmic drug loading.

DETAILED DESCRIPTION:
The purpose of this study is to determine if QT interval changes are detected during and after antiarrhythmic drug loading by the designed QT detection algorithm from LINQ ECG.

The QT intervals during the anti arrhythmic loading hospitalization period will be compared for all patients to analyze QT changes that may be caused due to antiarrhythmic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with LINQ/LINQII prior to the study enrollment (no more than 50% patients implanted with LINQII), but no greater than 2.5 years for LINQ or 3.5 years for LINQII, or patients who are indicated to receive a LINQ/LINQII implant at least 7 days prior to antiarrhythmic drug loading
* Patients who are scheduled to receive antiarrhythmic drug loading
* Age 18-80
* Patient is willing and able to comply with the protocol, including follow-up visits, and performing Holter recordings and patient activation transmissions

Exclusion Criteria:

* Patients who have a contraindication to long-term antiarrhythmic therapy
* Patients not suitable for long-term antiarrhythmic therapy
* Patients with a previous, existing cardiac implantation (i.e., cardiac pacemaker or cardiac resynchronization requiring > 40% pacing, implantable cardioverter defibrillator (ICDs))
* Patients with permanent and persistent AF
* Co-enrollment in another study or planning to participate in a concurrent device study during the course of this clinical study that could confound the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population for the LINQ QT Study is a patient implanted with LINQ/LINQII or scheduled for a LINQ/LINQII and who are scheduled to receive an antiarrhythmic drug loading, may undergo this study.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antony Chu, MD, Principal Investigator — Brown University
Locations (3):
- United States (3):
  - Baptist Hospital, Jacksonville, Florida
  - OhioHealth Research and Innovation Institute (OHRI), Columbus, Ohio
  - Bay Area Hospital, Coos Bay, Oregon

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual patient data with other researchers who were not investigators in the clinical study.

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: Anti-arrhythmic loading event
Period: Overall Study
Arm/Group | All Subjects
Started | 22
Completed | 18
Not Completed | 4
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Subjects with Completed Baseline and AA-loading Event
Groups:
- Subjects With Completed Baseline Anti Arrhythmic Loading Hospitalization: Characteristics of Subjects with completed Baseline Anti Arrhythmic Loading Hospitalization
Arm/Group | Subjects With Completed Baseline Anti Arrhythmic Loading Hospitalization
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 17
Age, Continuous [Mean (Full Range); unit: years] | 71.5 [40 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Medical History [Number; unit: participants]
  Transient Ischemic Attack | 1
  Thromboembolism | 1
  Stroke | 2
  Peripheral Artery Disease | 2
  Myocardial Infarction | 4
  Hypertension | 20
  Diabetes | 7
  Coronary Artery Disease | 8
  Congestive Heart Failure | 7
  Cancer | 1
  Aortic Plaque | 1
  Atrial Fibrillation | 21
  Atrial Flutter | 5

OUTCOME MEASURES:

1. Primary Outcome: QT Intervals During Antiarrhythmic Loading Hospitalization
Description: The QT intervals during antiarrhythmic loading will be compared for all patients with available LINQ ECG from the baseline anti arrhythmic loading hospitalization to analyze QT changes that may be caused due to antiarrhythmic drugs.
Time Frame: Assessed in the 2-hr period after each of the first four doses, difference between the maximum and minimum QTc interval reported
Population: 8 patients (avg. age 68±6.5 years, 63% males) with available LINQ ECG data during the anti arrhythmic loading hospitalization.
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- QTc Interval Trends Observed During the Anti Arrhythmic Loading Hospitalization: The maximum QTc interval in the 2-hr period after each of the first four anti arrhythmic doses.
Arm/Group | QTc Interval Trends Observed During the Anti Arrhythmic Loading Hospitalization
Number analyzed (Participants) | 8
milliseconds | 21.8 (9.4)

ADVERSE EVENTS:
Time Frame: 90 days
Groups:
- All Subjects: All Subjects Enrolled
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 1/21
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=21)
Hypokalemia (Renal and urinary disorders) | 1 (1)
Adverse Drug Reaction (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Continuous telemetered ICM ECG data available during the index antiarrhythmic loading hospitalization period was collected and available in 8 out of 21 patients enrolled (avg. age 68±6.5 years, 63% males) in the QT study and were included in this analysis. 12-lead ECG data was not available for 13 enrolled subjects due to Holter compatibility and technical issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol: LINQ QT Study Protocol (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT05488470/Prot_000.pdf